CLINICAL TRIAL: NCT02678949
Title: Changes in the Lung Clearance Index as Measured by Multiple-breath Washout, in Pediatric Patients With Asthma After Challenge With Inhaled Steroids and Short-acting Bronchodilator
Brief Title: Changes in the Lung Clearance Index in Pediatric Patients With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Jose Luis Lezana Fernandez, Pediatric Pulmonologist, Hospital Infantil de Mexico Federico Gomez
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HIMFG1
Record Dates: First submitted 2016-01-28; First posted 2016-02-10 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Childhood Asthma
MeSH Terms: interventions — Fluticasone; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inhaled Fluticasone 50 mcg/twice day (Experimental): Group 2; Inhaled fluticasone. 50 mcg/twice day for a period of 4 weeks.
  Interventions: Drug: Inhaled Fluticasone 50 mcg/twice day
- Inhaled Fluticasone 100 mcg/twice day (Experimental): Group 3;Inhaled fluticasone. 100 mcg/twice day for a period of 4 weeks
  Interventions: Drug: Inhaled Fluticasone 100 mcg/twice day
- Inhaled Albuterol (Experimental): Group 2 and group 3, inhaled albuterol one dose of 400 mcg.
  Interventions: Drug: Inhaled Albuterol

INTERVENTIONS:
Drug: Inhaled Fluticasone 50 mcg/twice day — After 7 days washout period, patients with mild asthma (group 2) will come to visit 2 where carried out a baseline spirometry and MBW test, subsequently will indicate them start treatment with inhaled fluticasone 50 mcg/twice a day, for a period of 4 weeks. At the end of the 4 weeks of treatment patients will come to Visit 3 and perform again spirometry and MBW test.
  Other Names: Fluticasone
  Arms: Inhaled Fluticasone 50 mcg/twice day
Drug: Inhaled Fluticasone 100 mcg/twice day — After 7 days washout period, patients with moderate asthma (group 3) will come to visit 2 where carried out a baseline spirometry and MBW test, subsequently will indicate them start treatment with inhaled fluticasone of 100 mcg/twice a day, for 4 weeks period. At the end of the 4 weeks of treatment patients will come to Visit 3 and perform again spirometry and MBW test.
  Other Names: Fluticasone
  Arms: Inhaled Fluticasone 100 mcg/twice day
Drug: Inhaled Albuterol — The patients in Group 2 and group 3 performing a baseline spirometry and MBW test, after which one dose of 400 mcg of inhaled albuterol will be administered. Twenty minutes after inhaling the dose of albuterol, spirometry and MBW test will be measured again in both groups.
  Other Names: Albuterol
  Arms: Inhaled Albuterol

SUMMARY:
The multiple breath washout (MBW) is one of pulmonary function test that displays flow and gas concentration plotted against time, and shows an exponential decay in end-tidal gas concentration (washout curve). A number of of indices to describe the washout curve have been proposed, the most commonly reported is the Lung Clearance Index (LCI). This is a simple measure of ventilation heterogeneity derived from MBW, that can be used after challenge with a short action bronchodilator and in response to inhaled steroids, both in the conductive airways as acinar. Patients with moderate and severe asthma are characterized by an abnormality in both, conductive and the acinar airway. Therefore the following research question could be: what are the abnormalities in the heterogeneity of ventilation in children with mild and moderate asthma, with respect to the healthy population measured by MBW, and whether these alterations persist after challenge with inhaled steroids and B2 agonists short-acting.

DETAILED DESCRIPTION:
The method most used to measure lung function, have been the spirometric tests, which generally reflect the function of the airway of highest caliber and elastic retraction of the lung. However, its use in clinical practice is limited by physiological variability and inconsistency in the measurements, therefore its value as a predictor of peripheral obstruction has been questioned. The Lung Clearance Index (LCI) is a simple measure of ventilation heterogeneity derived from multiple breath-washout (MBW) curve, that can be used after challenge with a short action bronchodilator and inhaled steroids, both in the conductive and acinar airways. Patients with moderate and severe asthma are characterized by an abnormality in both, conductive and the acinar airway. The LCI is one index derived from the concentration curves obtained during MBW to quantify the inefficiency in gas mixing of the lungs. A phase III slope analysis of the MBW curve can distinguish maldistribution of ventilation due to structural changes (acinar vs conductive lung zone). The conductive MBW index of ventilation heterogeneity is related to proximal lung structure, where convection dominates gas transport. The acinar MBW index of ventilation heterogeneity is related to peripheral lung, where convection-diffusion interaction occurs. Therefore the following research question could be: what are the abnormalities in the heterogeneity of ventilation in pediatric patients with a diagnosis of asthma, both mild and moderate, with respect to the healthy population, measured by MBW and whether these alterations persist using conventional treatment with inhaled steroids and B2 agonists short-acting.

The general objetive will be to identify changes in the LCI (heterogeneity of ventilation) retrieved from the MBW curve in children with diagnosis of mild and moderate asthma, before and after challenge with short-acting B2 agonists and after one month of treatment with knowledge dose of inhaled steroid.

Specific objectives;

1. . Difference in the baseline results of spirometry and LCI (derived form the MBW curve), between the control health group, and children with mild and moderate asthma.
2. . Changes in LCI (acinar or conductive ventilation heterogeneity) obtained from the MBW curve, from the baseline values and after challenge with short-acting B2 agonist and with inhaled steroids between groups of patients with mild or moderate asthma.
3. . Determine whether the alterations in the LCI of patients with mild and moderate asthma are originated from acinar or from the conductive airway.

Methodology. The LCI is calculated with the cumulative volume exhaled (CVE) during MBW test, divided between the functional residual capacity (FRC). This index is the number of turnovers of lung volume that the patient must breathe to clean the lungs of tracer gas (1/40th of the initial concentration). The expiratory N2 concentration will be plotted against volume changes between Total Lung Capacity (TLC) and Residual Volume (RV), and the slope (dN2) of the N2 alveolar plateau will be calculated by computer analysis of the best-fit line through phase III of the expiratory volume-concentration curve. The measurements will be accepted only if the vital capacity (VC) during the MBW is within 10% of the VC. During the MBW test, patients most perform a slow, full inspiratory and expiratory VC maneuver at inspiratory and expiratory flow rates of approximately 0.5 l/s.The VC will be obtained from the spirometry test.

Design; Clinical, controlled, parallel, longitudinal, comparative trial.

Sample universe; Patients of both sexes between 7-17 years of age that attending to Pediatric Pulmonology Service of the Hospital Infantil de Mexico, with a diagnosis of controlled mild or moderate asthma. It will included a control group (health children), as a criterion for normality and to compare the results of the spirometry and the LCI derived from the MBW curve obtained in this group, with the results of the same studies in a group of patients with mild and moderate asthma.

Inclusion criteria;

* For patients with asthma: Informed written consent signed by a parent or guardian of the patient and assent if signed by the patient.
* For control group: Informed written consent signed by parent or guardian consent and subject control where appropriate, signed by the subject.
* Patients from 7 to 17 years of age with a diagnosis of mild or moderate asthma according to the criteria of the Global Initiative for Asthma 2014 (Global Strategy for Asthma Management and Prevention. National Institutes of Health 2014), treated with inhaled steroids and who come to the outpatient clinic of Pediatric Pulmonology Service of Hospital Infantil de Mexico.
* An evolution of the asthma > 6 months.
* Control subjects (healthy) from 7 to 17, which will be contacted by telephone in accordance with a list that is counted in the Laboratory of Pulmonary Physiology who have participated in other studies or bioassays for calibration of equipment.
* Able to perform spirometry test and multiple-breath washout.
* No exacerbation of asthma in the past 4 weeks.
* Accept a washout period (without treatment) for 1 week before the realization of studies of pulmonary function (visit 2).
* Accept the use of short-acting B2 as necesary reason.
* Do not suffer from any other chronic disease, other than asthma.

Exclusion criteria;

* Patient with acute or chronic pulmonary disease other than asthma.
* Patient with a history of asthma exacerbation in the 4 weeks prior to inclusion in the study.
* Patients with a diagnosis of severe asthma according to criteria of the Global Initiative for Asthma 2014 (Global Strategy for Asthma Management and Prevention. National Institutes of Health 2014),
* Other co-morbidities.

Criteria of elimination;

* Patients who do not meet criteria of acceptability and repeatability at the spirometry, or MBW interpretation according with American Thoracic Society.
* Asthma exacerbation during the week of the washout period.
* Removal of informed consent.

Sample size; Taking into account the magnitude of the effect on the LCI during the MBW in pediatric subjects with asthma, pre and postbronchodilation on the basis of clinical studies carried out previously (Singer F, Abbas Ch, Yammine S, Casaulta C, Frey U, Latzin P. Abnormal small airway function in children with mild asthma.) Chest 2014; 145 (3): 492-499). Where the rate of LCI prebronchodilator was 2.96 ± 1.6 and the 20 minutes postbroncodilatador the clearance rate was 1.83 ± 1.24. Considering that the magnitude of the effect on the rate of LCI is 1.13, with standard deviation of 1.6. With a α = 0.05 (bilateral), β = 0.20, 80% statistical power. The sample size will be of 30 patients per group, taking into account a greater loss of 20%, the sample size will be increased to 35 subjects per group.

Selection of patients for the sample and its distribution; 3 groups of patients will be included: Group 1) Healthy group (controls). Group 2) Patients with mild asthma in treatment with low dose of inhaled steroids.

Group 3) Patients with moderate asthma in treatment with intermediatte dose of inhaled steroids.

Visit 1. Explanation of the study. Review of criteria for inclusion. Signature in the case of written informed consent. For Group 1; Only baseline spirometry and MBW test will be performed. No other intervention.

For groups 2 and 3. Be asked to suspend his current medication for 7 days (washout period), indicating only albuterol inhaled if necessary.

Visit 2 (1 week after Visit 1). Groups 2 and 3; baseline spirometry and MBW test. At the end of both studies, patients from to groups will receive one dose of 400 mcg of inhaled albuterol with spacer device. Twenty minutes after the dose of albuterol, they repeat spirometry and MBW test.

After patient have completed both studies, they will be asked to restart her medication with inhaled steroid; 100 mcg/day of fluticasone for the group of patients with mild asthma (Group 2) and 200 mcg/day of fluticasone for moderate asthma patients group (Group 3).

Visit 3 (4 weeks after Visit 2). Groups 2 and 3; basal spirometry and MBW test.

Statistical analysis. Descriptive statistics will by used to obtain measures of central tendency and dispersion in quantitative variables (average, standard deviation and 95% confidence interval). It will be compared and evaluate the effect of inhaled steroids and β2 agonists for short action on the rate of LCI and distribution of ventilation (acinar and conductive airways) through analysis of Student's t for related samples. The level of significance will be established with a p = ≤ 0.05.

Ethical Issues There will be any procedure until to obtain the approval of the Ethics Committee of the Hospital Infantil de México.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent signed by a parent or guardian of the patient and by the patient (asthma and healthy controls).
* Diagnosis of mild asthma and moderate asthma according to the criteria of the Global Initiative for Asthma 2014 (Global Strategy for Asthma Management and Prevention. National Institutes of Health 2014), treated with inhaled steroids and who come to the outpatient Clinic of Pediatric Pulmonology at Hospital Infantil de Mexico.
* An evolution of the asthma > 6 months.
* Able to perform spirometry test and multiple-breath washout test.
* No exacerbation of asthma in the past 4 weeks.
* Accept a washout period (without treatment) for 1 week before the realization of studies of pulmonary function.
* Accept the use of necessary short-acting B2 bronchodilator during the washout period.
* Do not suffer from any other chronic disease other than asthma.

Exclusion Criteria:

* Patient with acute or chronic pulmonary disease other than asthma.
* Patient with asthma exacerbation in the last 4 weeks prior to inclusion in the study.
* Patients with a diagnosis of severe asthma.
* Other co-morbidities.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effect of bronchodilator on the Lung Clearance Index between children with mild or moderate asthma | 20 minutes
  In all patients with asthma a multiple-breath washout (MBW) and standard spirometry will be perform before and after one dose of inhaled albuterol (400 mcg metered dose inhaler) delivered via standard spacer, in order to obtain forced expiratory volumen in 1 second (liters and percent of predicted value), functional residual capacity (FRC; liters and percent of predicted value) and Lung Clearance Index = cumulative expired volume/FRC.

SECONDARY OUTCOMES:
Change in the Lung Clearance Index after 4 weeks of treatment with inhaled fluticasone in children with mild asthma | 4 weeks
  Baseline spirometry and MBW for obtain the Lung Clearance Index conducted at visit 2 in children with mild asthma. After that, children will receive 50 mcg/twice a day, of inhaled Fluticasone for 1 month. At the end of 1 month of treatment, patients repeat spirometry and MBW in order to assess changes in the Lung Clearance Index
Change in the Lung Clearance Index after 4 weeks of treatment with inhaled fluticasone in children with moderate asthma | 4 weeks
  Baseline spirometry and MBW for obtain the Lung Clearance Index conducted at visit 2 in children with moderate asthma. After that, children will receive 100 mcg/twice a day of inhaled Fluticasone for 1 month. At the end of 1 month of treatment, patients repeat spirometry and MBW in order to assess changes in the Lung Clearance Index
Compare measures in the Lung Clearance Index betwwen children with and without asthma | 60 minutes
  Children in the healthy control group as well as children with mild or moderate asthma conducted a baseline standard spirometry and multiple-breath washout (MBW) in the first visit, according with the protocol and in order to obtain forced expiratory volumen in 1 second, functional residual capacity (FRC) and Lung Clearance Index = cumulative expired volume/FRC.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Lezana, MD, Principal Investigator — Hospital Infantil de Mexico Federico Gomez
Locations (1):
- Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Database

REFERENCES:
- [Background] Downie SR, Salome CM, Verbanck S, Thompson B, Berend N, King GG. Ventilation heterogeneity is a major determinant of airway hyperresponsiveness in asthma, independent of airway inflammation. Thorax. 2007 Aug;62(8):684-9. doi: 10.1136/thx.2006.069682. Epub 2007 Feb 20. PMID 17311839
- [Background] Martin RJ. Therapeutic significance of distal airway inflammation in asthma. J Allergy Clin Immunol. 2002 Feb;109(2 Suppl):S447-60. doi: 10.1067/mai.2002.121409. PMID 11842317
- [Background] Tulic MK, Christodoulopoulos P, Hamid Q. Small airway inflammation in asthma. Respir Res. 2001;2(6):333-9. doi: 10.1186/rr83. Epub 2001 Aug 10. PMID 11737932
- [Background] Enright PL, Lebowitz MD, Cockroft DW. Physiologic measures: pulmonary function tests. Asthma outcome. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 2):S9-18; discussion S19-20. doi: 10.1164/ajrccm/149.2_Pt_2.S9. PMID 8298772
- [Background] Ruppel GL, Enright PL. Pulmonary function testing. Respir Care. 2012 Jan;57(1):165-75. doi: 10.4187/respcare.01640. PMID 22222135
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Verbanck S, Schuermans D, Van Muylem A, Melot C, Noppen M, Vincken W, Paiva M. Conductive and acinar lung-zone contributions to ventilation inhomogeneity in COPD. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1573-7. doi: 10.1164/ajrccm.157.5.9710042. PMID 9603140
- [Background] Tashkin DP. The role of small airway inflammation in asthma. Allergy Asthma Proc. 2002 Jul-Aug;23(4):233-42. PMID 12221892
- [Background] Timmins SC, Diba C, Farrow CE, Schoeffel RE, Berend N, Salome CM, King GG. The relationship between airflow obstruction, emphysema extent, and small airways function in COPD. Chest. 2012 Aug;142(2):312-319. doi: 10.1378/chest.11-2169. PMID 22345381
- [Background] Verbanck S, Schuermans D, Paiva M, Vincken W. The functional benefit of anti-inflammatory aerosols in the lung periphery. J Allergy Clin Immunol. 2006 Aug;118(2):340-6. doi: 10.1016/j.jaci.2006.04.056. Epub 2006 Jun 21. PMID 16890756
- [Background] Verbanck S, Thompson BR, Schuermans D, Kalsi H, Biddiscombe M, Stuart-Andrews C, Hanon S, Van Muylem A, Paiva M, Vincken W, Usmani O. Ventilation heterogeneity in the acinar and conductive zones of the normal ageing lung. Thorax. 2012 Sep;67(9):789-95. doi: 10.1136/thoraxjnl-2011-201484. Epub 2012 Apr 27. PMID 22544894
- [Background] Macleod KA, Horsley AR, Bell NJ, Greening AP, Innes JA, Cunningham S. Ventilation heterogeneity in children with well controlled asthma with normal spirometry indicates residual airways disease. Thorax. 2009 Jan;64(1):33-7. doi: 10.1136/thx.2007.095018. Epub 2008 Aug 4. PMID 18678703
- [Background] Verbanck S, Schuermans D, Paiva M, Vincken W. Nonreversible conductive airway ventilation heterogeneity in mild asthma. J Appl Physiol (1985). 2003 Apr;94(4):1380-6. doi: 10.1152/japplphysiol.00588.2002. Epub 2002 Dec 6. PMID 12471044
- [Background] Verbanck S, Schuermans D, Vincken W. Inflammation and airway function in the lung periphery of patients with stable asthma. J Allergy Clin Immunol. 2010 Mar;125(3):611-6. doi: 10.1016/j.jaci.2009.10.053. Epub 2010 Feb 4. PMID 20132975
- [Background] Horsley A. Lung clearance index in the assessment of airways disease. Respir Med. 2009 Jun;103(6):793-9. doi: 10.1016/j.rmed.2009.01.025. Epub 2009 Feb 25. PMID 19246184
- [Background] Singer F, Abbas C, Yammine S, Casaulta C, Frey U, Latzin P. Abnormal small airways function in children with mild asthma. Chest. 2014 Mar 1;145(3):492-499. doi: 10.1378/chest.13-0784. PMID 24091465